CLINICAL TRIAL: NCT01005485
Title: Comprehensive Molecular and Morphologic Characterization of Circulating Endothelial Cells
Brief Title: Molecular and Morphologic Characterization of Circulating Endothelial Cells
Acronym: CEC
Status: Active, not recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute, Scripps Translational Science Institute
Other Study IDs: IRB#09-5287
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Myocardial Infarction (MI); Circulating Endothelial Cells (CEC); Control Group A: (Vascular Surgery); Control Group B: (Healthy controls)
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood for each patient will be collected from arterial access established as part of standard of care or via venipuncture. Blood must be collected in the order listed below. By drawing the PAX gene tube first, the likelihood of contamination of the sample with vessel wall endothelial cells is decreased.
  Enrollment:
  1. x 8.5 ml PAX gene (blue top) tube
  2. x 10 ml EDTA purple top tubes
  Follow-up visits: (healthy controls only)
  1. x 5 ml red top (discard)
  2. x 10 ml EDTA purple top tube
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Patients undergoing open vascular surgery on arterial structures to better define optimal laboratory and collection techniques for isolation of CECs.
- Group B: Healthy controls will be recruited from the general medical population, community.
- Acute Myocardial Infarction: Patients with acute myocardial infarction with or without ST segment deviation.

SUMMARY:
The primary hypothesis of this study is that circulating endothelial cells (CECs) harbor key genetic and structural characteristics predisposing individuals to acute atherosclerotic plaque rupture and heart attack.

DETAILED DESCRIPTION:
Endothelial injury and inflammation are pivotal underlying processes that put patients at risk for catastrophic vascular events including acute myocardial infarction (heart attack) and stroke. We seek to accelerate scientific discovery through clinically meaningful, innovative translational research, and are collaborating in a trans-disciplinary effort to define the DNA sequence of CECs and that of germ line DNA, along with RNA sequencing, mRNA expression profiling, and ultrastructural characterization of CECs in order to better understand the mechanisms leading to acute arterial plaque rupture and embolization of arterial endothelial cells in patients with acute myocardial infarction. This will enable us to create a molecular fingerprint that could identify and preempt individuals from suffering from such debilitating vascular conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80 years old.
2. Must be reliable, cooperative and willing to comply with all protocol-specified procedures if consented.
3. Able to understand and grant informed consent
4. Subjects must meet one of the following (a-c):

   1. Healthy control subjects not meeting any exclusion criteria for controls below
   2. Patients scheduled for an open vascular procedure of an arterial structure
   3. Patients with acute MI defined as:

   i. Clinical history and symptoms consistent with acute MI AND ii Elevated cardiac markers (CKMB, Troponin I or T) consistent with MI (abnormals are according to enrolling institution's lab standards) AND iii. Able to complete study enrollment (consent & blood draw) within 48 hours of presentation to the study site.

Exclusion Criteria:

General Exclusion Criteria:

1. Has a significant medical condition that in the investigator's opinion may interfere with the patient's optimal participation in the study.

Exclusion for Healthy Controls:

1. Age greater than 35
2. Previous history of coronary artery disease or MI
3. Diabetes
4. Peripheral arterial disease
5. Hypertension (>140/90 or on blood pressure medication)
6. Sickle cell disease
7. Acute or Chronic kidney disease
8. Acute or Chronic vascular conditions, not otherwise specified
9. Active or history of inflammation of connective tissue and vascular structures (i.e. vasculitis, rheumatoid arthritis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the general in-patient and out-patient populations for myocardial infarction and/or vascular surgery. Healthy controls will be recruited from the general medical population and community.
Sampling Method: Non-Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2010-01; Primary Completion 2017-04 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is complete molecular profiling of CEC's in up to 250 patients with a diagnosis of acute myocardial infarction (MI) and up to 25 healthy controls. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Topol, M.D., Principal Investigator — Scripps Translational Science Institute
Locations (1):
- Scrippshealth, La Jolla, California, United States